CLINICAL TRIAL: NCT03829566
Title: Autologous Hematopoietic Stem Cell Transplant for Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Autologous Transplant To End NMO Spectrum Disorder
Acronym: ATTEND
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Discontinued by Investigator
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD.ATTEND.2018
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Neuromyelitis Optica; Devic's Disease; NMO Spectrum Disorder
Keywords: Autologous Stem Cell Transplantation; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Rituximab; Cyclophosphamide; Mesna; thymoglobulin; Antilymphocyte Serum; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Granulocyte Colony-Stimulating Factor; Filgrastim; Immunoglobulins, Intravenous; Immunoglobulin G; Octagam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with rituximab, cyclophosphamide, mesna, rATG (rabbit), and methylprednisolone. Granulocyte-colony stimulating factor (G-CSF) and intravenous immunoglobulin (IVIg) will be administered post-transplant.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: G-CSF; Biological: IVIg; Biological: Autologous Stem Cells

INTERVENTIONS:
Drug: Rituximab — Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Other Names: Rituxan
Drug: Cyclophosphamide — A medication used as chemotherapy and to suppress the immune system
  Other Names: Cytoxan
Drug: Mesna — A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  Other Names: Mesnex
Drug: rATG — A rabbit polyclonal antibody to lymphocytes
  Other Names: Thymoglobulin; Anti-Thymocyte Globulin
Drug: Methylprednisolone — A corticosteroid medication used to suppress the immune system and decrease inflammation
  Other Names: Solu-Medrol; Depo-Medrol
Drug: G-CSF — A glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; Filgrastim; Granix; Zarxio
Biological: IVIg — Pooled immunoglobulin (IgG) from thousands of plasma donors that has immunomodulatory and anti-inflammatory effects
  Other Names: Bivigam; Carimune Nanofiltered (NF); Gammagard; Privigen; Octagam
Biological: Autologous Stem Cells — Infusion of patient's own stem cells

SUMMARY:
This study is designed to treat your disease with an autologous stem cell transplant using a regimen of immune suppressant drugs and chemotherapy to reset your immune system and to determine if your disease will go into long-term remission.

DETAILED DESCRIPTION:
The autologous stem cell transplant used in this research study is an investigational procedure that uses cyclophosphamide (chemotherapy), rabbit antithymocyte globulin (rATG) (a protein that kills the immune cells that are thought to be causing your disease), rituximab (a biologic drug that targets B cells of your immune system), and intravenous immunoglobulin (IVIg) (pooled IgG antibodies from plasma donors with immunomodulatory and anti-inflammatory effects), followed by return of your own previously collected blood stem cells (autologous stem cell transplant). One day of plasmapheresis will also be performed the day prior to admission for stem cell transplant to remove disease-causing antibodies. The ability of this experimental treatment to stop relapses and progression (worsening) of your NMOSD will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 years old at the time of pre-transplant evaluation
2. An established diagnosis of NMOSD (with or without aquaporin 4 (AQP4)-IgG antibody)

Exclusion Criteria:

1. Under age of 18 or over age of 65
2. Prisoners
3. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible, or any adult who is unable to consent (for adults cognitively impaired due to disease, consent may be obtained from the closest living relative).
4. Paraplegia or quadriplegia (must be able to use a walker if even for only a few feet)
5. Extensive subcortical white matter lesions
6. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment
7. Myocardial infarction within the last 12 months. If longer than 12 months, must pass a dobutamine stress test and be cleared by cardiology.
8. Active systemic lupus erythematous, Sjogren's, myasthenia gravis, or another autoimmune disease
9. Sickle cell disease, sickle cell disease, or coagulopathy
10. Prior history of malignancy that required any radiotherapy, chemotherapy, or biological therapy
11. Positive pregnancy test, inability or unable to pursue effective means of birth control, or failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
12. Women who are breastfeeding
13. Untreated life-threatening cardiac arrhythmia on electrocardiogram (EKG) or 24-hour holter
14. Left ventricular ejection fraction (LVEF) <50%
15. Tiffeneau-Pinelli index (FEV1/FVC) <70% of predicted after bronchodilator therapy (if necessary), or diffusing capacity of lung for carbon monoxide (DLCO) hemoglobin corrected <70 % predicted
16. Serum creatinine >2.0 mg/dl
17. Liver cirrhosis, transaminases >2x of normal limits, or bilirubin >2.0 mg/dl unless due to Gilbert's disease
18. Major hematological abnormalities such as platelet count < 100,000/μl or absolute neutrophil count (ANC) < 1000/μl
19. Active infection except asymptomatic bacteriuria
20. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have magnetic resonance imaging (MRI) exams
21. Known hypersensitivity to mouse, rabbit, or E. coli derived proteins
22. Human immunodeficiency virus (HIV) positive
23. Hepatitis B or C positive
24. Use of natalizumab (Tysabri) within the previous six months
25. Use of fingolimod (Gilenya) within the previous three months
26. Use of dimethyl fumarate (Tecfidera) within the previous three months
27. Use of teriflunomide (Aubagio) unless cleared from the body (plasma concentration <0.02mcg/ml) following elimination from the body with cholestyramine 8g three times a day for 11 days
28. Use of alemtuzumab (Lemtrada/Campath) within previous 12 months
29. Use of rituximab (Rituxan) or ocrelizumab (Ocrevus) within previous six months
30. Prior treatment with mitoxantrone (Novantrone)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 5 years
  Disease progression defined as: 1.0-point increase in the Expanded Disability Status Scale (EDSS) on consecutive evaluations at least six months apart and not due to a non-NMO disease process. The EDSS scale ranges from 0 to 10 in 0.5 increments that represent higher levels of disability.

SECONDARY OUTCOMES:
Relapse-Free Survival | 5 years
  Relapse defined as: Acute neurologic deterioration occurring after engraftment and lasting more than 24 hours, accompanied by objective worsening on neurological examination that are documented by a neurologist and not explained by fever, infection, stress, heat, drugs or related pseudo-exacerbation. Supportive confirmation by enhancement on MRI is preferred but not mandatory.
Expanded Disability Status Scale (EDSS) Improvement | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The EDSS scale ranges from 0 to 10 in 0.5 increments that represent higher levels of disability. Improvement in EDSS is defined by both a 0.5 or 1.0 points sustained for more than 6 months
Scripps Neurological Rating Scale (NRS) Improvement | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The NRS scale ranges from 0 to 100 in 1 point increments that represent lower levels of disability.
Improvement in Quality of Life | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Measured using the short form (SF)-36 health survey.
Paced Auditory Serial Addition Test (PASAT) Improvement | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Improvement measured with the 2" and 3" versions
Ambulation Index Improvement | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The subject's walk of 25 feet is timed and a score from 0 to 10 is assigned based on their walk/gait and/or assistance required.
9 Hole Peg Test (9-HPT) Improvement | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The 9-HPT is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice, with the total time to complete the task each time recorded and then averaged.
Change in NMO IgG (aquaporin-4) Antibody Titer | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Evaluation of the antibody titer, looking for a change from positive to negative.
Improvement in Visual Acuity | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  A visual acuity test is an eye exam that checks how well one sees the details of a letter or symbol from a specific distance.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No